CLINICAL TRIAL: NCT01536665
Title: The Effect of Liraglutide Adjunct to Insulin on Glucagon Response to Hypoglycaemia in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9211-3953; U1111-1123-9882 (Other: WHO); 2011-004240-22 (EudraCT Number)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- Medium (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- High (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Administered subcutaneously (s.c., under the skin) once daily for 4 weeks.
Drug: placebo — Administered subcutaneously (s.c., under the skin) once daily for 4 weeks.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate if liraglutide adjunct to insulin treatment changes the glucagon response during hypoglycaemia in subjects with type 1 diabetes compared with conventional insulin treatment after 4 weeks' treatment with liraglutide or placebo.

Subjects will initially be randomised to one of the three dose groups, and subsequently randomly allocated to one of two treatment sequences (liraglutide/placebo or placebo/liraglutide).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months prior to randomisation
* Body mass index (BMI) between 20.0 and 28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Use of liraglutide or exenatide within 3 months of randomisation
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the trial physician or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Geometric mean glucagon concentration during hypoglycaemia (nadir glucose (target 2.5 mmol/L) ) | At week 4

SECONDARY OUTCOMES:
Geometric mean glucagon concentration at plasma glucose levels other than nadir | At week 4
Geometric mean concentrations of adrenaline and noradrenaline at nadir | At week 4
Time from termination of insulin infusion at nadir to reach plasma glucose 4.0 | At week 4

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Result] Mader JK, Jensen L, Ingwersen SH, Christiansen E, Heller S, Pieber TR. Pharmacokinetic Properties of Liraglutide as Adjunct to Insulin in Subjects with Type 1 Diabetes Mellitus. Clin Pharmacokinet. 2016 Nov;55(11):1457-1463. doi: 10.1007/s40262-016-0413-4. PMID 27282158
- [Result] Pieber TR, Deller S, Korsatko S, Jensen L, Christiansen E, Madsen J, Heller SR. Counter-regulatory hormone responses to hypoglycaemia in people with type 1 diabetes after 4 weeks of treatment with liraglutide adjunct to insulin: a randomized, placebo-controlled, double-blind, crossover trial. Diabetes Obes Metab. 2015 Aug;17(8):742-50. doi: 10.1111/dom.12473. Epub 2015 May 20. PMID 25855340
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com